CLINICAL TRIAL: NCT04287309
Title: CAR-T Cellular Therapy for B Cell Malignancies Involved in Central Nervous System
Brief Title: CAR-T Cellular Therapy for B Cell Malignancies Involved in CNS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, He Huang, Professor, Zhejiang University
Other Study IDs: 19-002
Record Dates: First submitted 2020-02-22; First posted 2020-02-27 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Hematological Malignancy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood and cerebral fluid for CAR-T cell expansion, serum for cytokine concerntraion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CAR-T cells — CD19 targeted CAR-T treatment

SUMMARY:
This is a single arm, open-label, single-center study. This study is indicated for relapsed or refractory CD19+ B-line hematological malignancy involved in CNS. 20 patients were enrolled. Primary objective is to explore the safety. The secondary objective is to explore the efficacy.

DETAILED DESCRIPTION:
This is a single arm, open-label, single-center study. This study is indicated for relapsed or refractory CD19+ B-line hematological malignancy involved in CNS. All together 20 patients were enrolled. Primary objective is to explore the safety including the complication of cytokine release syndrome, CRES, pancytopenia and infection. The secondary objective is to explore the efficacy. We will also detect CAR-T cell expansion dynamics in blood and cerebral fluid and compare the difference.

ELIGIBILITY:
Inclusion Criteria:

1.Male or female aged ≥ 3 and <70 years old; 2.Histologically confirmed diagnosis of CD19+ B cell malignancies involved in CNS 3.Relapsed or refractory CD19+ B cell malignancies 4.total bilirubin ≤ 51umol/L, ALT and AST ≤ 3 times of upper limit of normal, creatinine ≤ 176.8umol/L; 5.Echocardiogram shows left ventricular ejection fraction (LVEF) ≥ 50%; 6.No active infection in the lungs, blood oxygen saturation by sucking air is ≥ 92%; 7.Estimated survival time ≥ 3 months; 8.ECOG performance status 0 to 2; 8.Patients or their legal guardians volunteer to participate in the study and sign the informed consent.

Exclusion Criteria:

1. Patients with hereditary syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome or any other known bone marrow failure syndrome;
2. extensive involvement of gastrointestinal lymphoma;
3. radiotherapy, chemotherapy and monoclonal antibody within 1 week before screening;
4. Have a history of allergy to any of the components in the cell products;
5. According to the New York heart association (NYHA) cardiac function classification criteria, Subjects with grade III or IV cardiac insufficiency;
6. Myocardial infarction, cardioangioplasty or stenting, unstable angina pectoris, or other severe cardiac diseases within 12 months of enrollment;
7. Severe primary or secondary hypertension of grade 3 or above (WHO Hypertension Guidelines, 1999);
8. Electrocardiogram shows prolonged QT interval, severe heart diseases such as severe arrhythmia in the past;
9. Patients with severe active infections (excluding simple urinary tract infection and bacterial pharyngitis).
10. Indwelling catheters in vivo (e.g. percutaneous nephrostomy, Foley catheter, bile duct catheter, or pleural/peritoneal/pericardial catheter). Ommaya storage, dedicated central venous access catheters such as Port-a-Cath or Hickman catheters are allowed;
11. History of other primary cancer, except for the following conditions:

    1. Cured non-melanoma after resection, such as basal cell carcinoma of the skin;
    2. Cervical cancer in situ, localized prostate cancer, ductal cancer in situ with disease-free survival ≥ 2 years after adequate treatment;
12. Patients with graft-versus-host disease (GVHD);

19.Prior immunizations with live vaccine 4 weeks prior to screening; 13.History of alcoholism, drug abuse or mental illness; 14.Concurrent therapy with systemic steroids within 1 week prior to screening, except for the patients recently or currently receiving inhaled steroids; 15.Patients who have participated in any other clinical studies within 2 weeks prior to screening; 16.pregnant and breast-feeding women and the subjects who are fertile and unable to take effective contraceptive measures (regardless of the gender); 17.Any situations that the investigator believes may increase the risk of patients or interfere with the results of study.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CNS involvement
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-02-28 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Adverse events that related to treatment | 2 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)

SECONDARY OUTCOMES:
The response rate of CAR-T treatment in patients with relapse/refractory B cell malignancies involved in CNS that treated by CD19 CAR-T cells therapy | 6 months
  The response rate of BCMA CAR-T treatment will be recorded and assessed according to WHO criteria

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Hospital of Zhejiang Medical Colleage Zhejiang University, Hangzhou, Zhejiang
  - the First Affiliated Hospital,School of Medicine, Zhejiang University, Hangzhou, Zhejiang